CLINICAL TRIAL: NCT04744350
Title: Conservative or Operative Therapy in Patients With a Fragility Fracture of the Pelvis: a Prospective, Randomized Controlled Trial
Brief Title: Conservative or Operative Therapy in Patients With a Fragility Fracture of the Pelvis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Björn-Christian Link (Other)
Responsible Party: Sponsor-Investigator, Björn-Christian Link, Co-director of the orthopaedics and traumatology department, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFP1
Record Dates: First submitted 2020-12-10; First posted 2021-02-08 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Active Comparator): Surgical treatment using a minimal invasive surgical method. At our hospital we perform a percutaneous sacroiliac osteosynthesis using cannulated, perforated and fenestrated screws. This procedure is preferably performed in our hybrid operation theatre, which allows for correct placement using an intraoperative CT-scan.
  Interventions: Procedure: Treatment of FFP type IIb and IIc
- Conservative (Active Comparator): Patients will receive individually tailored physiotherapy and analgesics if necessary.
  Interventions: Procedure: Treatment of FFP type IIb and IIc

INTERVENTIONS:
Procedure: Treatment of FFP type IIb and IIc — Patients will either be randomized in the surgical or conservative group.

SUMMARY:
In our society the population consists of more elderly patients. Medical treatment needs to be adjusted to this patient group. This research project focusses on patients with a fragility fracture of the pelvis. This results from a minor trauma and can cause a long immobilization period because of severe pain. For FFP type II b and II c there is no consensus on the best treatment option. Either a surgical minimal invasive sacroiliac osteosynthesis or conservative treatment is a possibility. Of course, both treatment options have pros and cons. This research project will randomize all patients with a FFP IIb or IIc fracture in either surgical or conservative treatment. These treatments will be evaluated at the follow-ups, 4 weeks, 4 months and 1 year after trauma. This will be evaluated with the DEMMI, Accelerometer, EQ-5D (EuroQol Quality of Live Questionnaire), radiological results, range of motion, pain-levels and reporting any postoperative complications or adverse events. Patient will be included over a period of 18 months and will be followed for at least a year. This research project aim to answer the question which treatment option for FFP type IIb and IIc is the most adequate.

DETAILED DESCRIPTION:
Background. Fragility fractures of the pelvis are increasing in incidence. These are osteoporotic fractures, who result from a minor trauma. Typically, the weak osteoporotic bone is fractured, an the ligaments remain intact resulting in an undisplaced or minimally displaced pelvic ring. Fragility fractures of the pelvis can be divided in type I, II, III and IV. For type I the treatment method of choice is conservative. For type III and IV a surgical treatment is necessary. Only the ideal treatment for type II remains unclear. There is no consensus in whether conservative treatment or surgical treatment will have the best outcomes. Surgical treatment mostly means a minimal invasive osteosynthesis. In our hospital we use percutaneous sacroiliac screw fixation with augmentation. The screws used are perforated and fenestrated, allowing for a correct placement an cement augmentation. Preferably, this procedure is performed in our hybrid operation theatre. An intraoperative CT-scan can be performed. This treatment method has proven to be a safe method in literature. On the other hand, surgical treatment, can have complications and risks, especially in the elderly. Conservative treatment consist of mobilisation and physiotherapy. But conservative treatment can be limited because of uncontrolled pain, resulting in a long immobilisation period. Immobilisation in the elderly leads to several complications. This research project will focus on early operative intervention to reduce the immobilisation period and its negative consequences.

Study design. Recruitment of patients will find place in our emergency department and our outpatient clinic. A lot of patients with a FFP type IIb and IIc present themselves at our emergency department due to immobilising pain. All the elderly patient who complain about sacroiliac pain will receive an CT-scan. Literature showed that an conventional x-ray is not sufficient to detect sacroiliac fractures. On the other hand a lot of patient are referred to our outpatient clinic by other hospitals in our region or even general practioners. All these patients, who meet our inclusion criteria, will be asked for informed consent. After informed consent has been collected, patients will be randomised to on of the groups. The first group will receive surgical treatment and the second group will receive conservative treatment. Randomisation is performed with a vending machine. Depending on which soda can comes out, patients are assigned to the groups.

Study intervention. As stated before the are two groups in this research project. Both treatment are standard treatments. Both groups will receive a standard set of co-interventions, such as adequate analgesics and intensive physiotherapy. At our hospital a geriatric trauma centre is established. After discharge or 4 weeks after trauma a first follow-up is planned. This is primary for the treatment evaluation. Then after 4 months are second follow-up is planned with a traumatologist, physiotherapist and a geriatric specialist. At this follow-up several benchmark test are performed, such as the DEMMI, EQ 5D and an accelerometer is explained and given out. Especially this accelerometer will tell us more about the amount of mobilisation or immobilisation at home. The last follow-up will be 1 year after trauma. At all follow-ups radiological controls are performed. These will be conventional x-rays. Only in specific cases, for example prolonged pain, an CT-scan will be performed.

Data and data management. The sample size was based on the expected difference between treatment groups in improvement on the DEMMI score between baseline and 4 months follow-up. Previous studies show that the minimal clinical important difference of the DEMMI score is 10 points. This results in a sample size of 68 patients, accounted for 10% loss to follow-up.

The statistical planned analyses are primary a pearson chi-squared or fishers exact test for categorical variables or a students t or mann-whitney test. However the primary outcome will be analysed using mixed linear models with random effects. The models will be compared usin Akaike information criterium. Missing data will be imputed using multiple imputation. All analyses will be performed using SPSS version 19 or higher. A p value <0.05 is regarded as being statistically significant.

Data is stored on the protected server systems of Hospital of Lucerne. Files containing anonymous data can also be stored on the personal computers of the investigators. Data is recorded on paper and digitally. Questionnaires are on paper, but all the measurements, as the DEMMI score of range of motion will be digitally. Participants can not be identified in the CRF (Case report form). Appropriate corresponding codes are only known and accessible for the investigators.

Upon simple request by the patient, he or she will immediately be withdrawn from the study and no further date will be recorded in the study. It is guaranteed that further treatment will be equal to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* The fracture must be a fragility fracture. This means absence of high energy trauma.
* Fragility fracture of the sacrum (FFP II b + c). Involvement of the ventral pelvic ring is not an exclusion criteria.
* Able to walk 4 meters before fracture

Exclusion Criteria:

* Patients who had a high energy trauma.
* FFP I or FFP III+IV were operative therapy is recommended
* Patient who are not operable according to the anaesthesiologist on call.
* Open fractures.
* Revision surgeries.
* Absent contact information
* Living abroad and cannot participate in follow-up visits.
* Withdrawal from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mobility level | 1 year
  DEMMI (0-100, 100 is maximal mobility)

SECONDARY OUTCOMES:
Pain levels | 1 year
  VAS (visual analogue scale, 0-10, 0 means no pain)
Clinical characteristics | Baseline
  Age
Clinical characteristics | Baseline
  Gender
Clinical characteristics | Baseline
  ASA-Score (1-6, 1 is a healthy patient)
Clinical characteristics | Baseline, 1 year
  BMI
Clinical characteristics | Baseline
  Osteoporosis treatment (yes or no)
Medication | Baseline, 1 year
  Reporting what kind of medications all patients take (including steroids, anticoagulation, pain killers, et cetera)
Clinical characteristics | Through study completion, an average of 1 year
  Surgical related complications
Clinical characteristics | after discharge
  Length of hospital stay after first admission
Clinical characteristics | Baseline
  Fracture classification (FFP I - IV)
Clinical characteristics | 1 year
  FES-1 (falls efficacy scale, 16-64, 16 means no fear of falling, 64 is the maximum)
Clinical characteristics | 1 year
  EQ-5D (0-100, 100 is the best possible health status)
Clinical characteristics | 1 year
  SPPB (short physical performance battery, 0-12, 12 is the best function)
Mobility level | 1 year
  Barthel Index (0-100, 100 is completely independent)
Mobility level | During 1 week after 4 Months
  Accelerometer (this is a device that continously measures the activity level of an patient. It comes in the form of a bracelet)
Mobility level | 1 year
  TUG (time up and go test)
Mobility level | 1 year
  5 Chair rise

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oberkircher L, Ruchholtz S, Rommens PM, Hofmann A, Bucking B, Kruger A. Osteoporotic Pelvic Fractures. Dtsch Arztebl Int. 2018 Feb 2;115(5):70-80. doi: 10.3238/arztebl.2018.0070. PMID 29439771
- [Background] Fuchs T, Rottbeck U, Hofbauer V, Raschke M, Stange R. [Pelvic ring fractures in the elderly. Underestimated osteoporotic fracture]. Unfallchirurg. 2011 Aug;114(8):663-70. doi: 10.1007/s00113-011-2020-z. German. PMID 21800137
- [Background] Rommens PM, Wagner D, Hofmann A. [Osteoporotic fractures of the pelvic ring]. Z Orthop Unfall. 2012 Jun;150(3):e107-18; quiz e119-20. doi: 10.1055/s-0032-1314948. Epub 2012 Jun 21. German. PMID 22723074
- [Background] Rommens PM, Hofmann A. Comprehensive classification of fragility fractures of the pelvic ring: Recommendations for surgical treatment. Injury. 2013 Dec;44(12):1733-44. doi: 10.1016/j.injury.2013.06.023. Epub 2013 Jul 18. PMID 23871193
- [Background] Matta JM, Saucedo T. Internal fixation of pelvic ring fractures. Clin Orthop Relat Res. 1989 May;(242):83-97. PMID 2706863
- [Background] Rommens PM, Wagner D, Hofmann A. Minimal Invasive Surgical Treatment of Fragility Fractures of the Pelvis. Chirurgia (Bucur). 2017 Sept-Oct;112(5):524-537. doi: 10.21614/chirurgia.112.5.524. PMID 29088552
- [Background] Richter PH, Gebhard F, Dehner C, Scola A. Accuracy of computer-assisted iliosacral screw placement using a hybrid operating room. Injury. 2016 Feb;47(2):402-7. doi: 10.1016/j.injury.2015.11.023. Epub 2015 Dec 12. PMID 26708797
- [Background] Wahnert D, Raschke MJ, Fuchs T. Cement augmentation of the navigated iliosacral screw in the treatment of insufficiency fractures of the sacrum: a new method using modified implants. Int Orthop. 2013 Jun;37(6):1147-50. doi: 10.1007/s00264-013-1875-8. Epub 2013 Apr 4. PMID 23553117
- [Background] Routt ML Jr, Simonian PT, Mills WJ. Iliosacral screw fixation: early complications of the percutaneous technique. J Orthop Trauma. 1997 Nov;11(8):584-9. doi: 10.1097/00005131-199711000-00007. PMID 9415865
- [Background] Konig MA, Hediger S, Schmitt JW, Jentzsch T, Sprengel K, Werner CML. In-screw cement augmentation for iliosacral screw fixation in posterior ring pathologies with insufficient bone stock. Eur J Trauma Emerg Surg. 2018 Apr;44(2):203-210. doi: 10.1007/s00068-016-0681-6. Epub 2016 May 11. PMID 27167237
- [Background] Wagner D, Ossendorf C, Gruszka D, Hofmann A, Rommens PM. Fragility fractures of the sacrum: how to identify and when to treat surgically? Eur J Trauma Emerg Surg. 2015 Aug;41(4):349-62. doi: 10.1007/s00068-015-0530-z. Epub 2015 Apr 18. PMID 26038048
- [Background] Hopf JC, Krieglstein CF, Muller LP, Koslowsky TC. Percutaneous iliosacral screw fixation after osteoporotic posterior ring fractures of the pelvis reduces pain significantly in elderly patients. Injury. 2015 Aug;46(8):1631-6. doi: 10.1016/j.injury.2015.04.036. Epub 2015 May 14. PMID 26052052
- [Background] Konig A, Oberkircher L, Beeres FJP, Babst R, Ruchholtz S, Link BC. Cement augmentation of sacroiliac screws in fragility fractures of the pelvic ring-A synopsis and systematic review of the current literature. Injury. 2019 Aug;50(8):1411-1417. doi: 10.1016/j.injury.2019.06.025. Epub 2019 Jun 28. PMID 31301810
- [Background] Hobart JC, Thompson AJ. The five item Barthel index. J Neurol Neurosurg Psychiatry. 2001 Aug;71(2):225-30. doi: 10.1136/jnnp.71.2.225. PMID 11459898
- [Background] de Morton NA, Davidson M, Keating JL. The de Morton Mobility Index (DEMMI): an essential health index for an ageing world. Health Qual Life Outcomes. 2008 Aug 19;6:63. doi: 10.1186/1477-7525-6-63. PMID 18713451
- [Background] Ruhle A, Oehme F, Link BC, Metzger J, Fischer H, Stickel M, Delagrammaticas DE, Babst R, Beeres FJP. Swiss chocolate and free beverages to increase the motivation for scientific work amongst residents: a prospective interventional study in a non-academic teaching hospital in Switzerland. Trials. 2020 Jan 13;21(1):74. doi: 10.1186/s13063-019-3956-5. PMID 31931852
- [Background] Unnanuntana A, Laohaprasitiporn P, Jarusriwanna A. Effect of bisphosphonate initiation at week 2 versus week 12 on short-term functional recovery after femoral neck fracture: a randomized controlled trial. Arch Osteoporos. 2017 Dec;12(1):27. doi: 10.1007/s11657-017-0321-8. Epub 2017 Mar 10. PMID 28283937
- [Derived] Haveman RA, van de Wall BJM, Rohner M, Beeres FJP, Haefeli PC, Baumgartner R, Babst R, Link BC. Conservative or operative therapy in patients with a fragility fracture of the pelvis: study protocol for a prospective, randomized controlled trial. Trials. 2024 Jul 30;25(1):513. doi: 10.1186/s13063-024-08350-z. PMID 39080698